CLINICAL TRIAL: NCT05325827
Title: Effect of Ultrasound-guided High Fascia Iliaca Compartment Block in Patients Undergoing Arthroscopic Knee Surgery: A Prospective, Double-Blind, Randomized, Clinical Trial
Brief Title: Effect of Ultrasound-guided H-FICB in Patients Undergoing Arthroscopic Knee Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Affiliated Hospital of Nantong University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2022-K022
Record Dates: First submitted 2022-04-06; First posted 2022-04-13 (Actual); Last update posted 2022-04-13 (Actual); Status verified 2022-04

CONDITIONS: Knee Disease; Delirium
MeSH Terms: conditions — Delirium

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A: H-FICB under ultrasound guidance before general anesthesia (Experimental): Group A was subjected to a high fascia iliaca compartment block under ultrasound guidance before general anesthesia.
  Interventions: Procedure: ultrasound-guided high fascia iliaca compartment block
- Group B: FBC combined with SBC under ultrasound guidance before general anesthesia (No Intervention): Group B was subjected to a femoral nerve block combined with a sciatic nerve block under ultrasound guidance before general anesthesia.

INTERVENTIONS:
Procedure: ultrasound-guided high fascia iliaca compartment block — H-FICB was guided by ultrasound before general anesthesia. The patient was supine. First, the probe is placed transversely above the groin. Then slide the probe up and down to reveal a clear image of the internal oblique and sartorius muscles. There is a bowtie-like iliac fascia space at the junction of these two muscles. After the scanning, the needle was inserted behind the probe with the tip pointed to the ventral side under the guidance of real-time ultrasound; the tip passed through the skin into the iliac fascia space and advanced to the inguinal ligament. After no blood was extracted, 1 ~ 2 ml of normal saline was firstly injected to determine whether the tip position was correct. If the needle tip was correctly positioned, 0.375% ropivacaine 30 mL of local anesthetic was injected. The H-FICB was performed under ultrasound guidance by the same anesthesiologist.
  Arms: Group A: H-FICB under ultrasound guidance before general anesthesia

SUMMARY:
Arthroscopic knee surgery is a minimally invasive operation. Postoperative pain usually occurs, especially within 24 hours after surgery, the incidence of pain can be more than 76%. Pain will affect the patient's emotions and life, cause adverse effects, and even lead to postoperative delirium. This study aimed to investigate the clinical effect of ultrasound-guided high fascia iliaca compartment block(H-FICB) in patients undergoing knee arthroscopy and to compare it with the normal method which is femoral nerve block combined with a sciatic nerve block to choose the better way. A double-blind, randomized controlled trial was conducted with 44 patients, aged 18-65 years, ASA I-III, who were scheduled to undergo arthroscopic knee surgery in our hospital were selected, the patients were divided into Group A and Group B by random number table method, with 22 patients in each group. Group A was subjected to the H-FICB under ultrasound guidance before general anesthesia, given 0.375% ropivacaine 30 ml. Group B received ultrasound-guided femoral nerve block combined with sciatic nerve block before general anesthesia, given 0.375% ropivacaine 30 ml.

The mini-mental State Examination was used to assess all the patients' primary cognitive status one day before surgery. The initial acting time and the degrees of sensory block and motor block were recorded after the nerve block was completed. Perioperative variables were recorded to be compared. The investigators used the visual analog scale to assess patients' pain degree with postoperative, recorded the occurrence of adverse events such as postoperative nausea and vomiting(PONV), delayed emergence from anesthesia, and respiratory depression. The confusion assessment method was used to assess whether patients experienced delirium.

DETAILED DESCRIPTION:
1. Study design and setting 44 patients undergoing arthroscopic knee surgery under general anesthesia, gender, aged 18-65 years, American Society of Anesthesiologists (ASA) physical status I-III. Exclusion criteria: MMSE of 1 day before surgery < 27, communication and dysfunction (e.g., vision, hearing), cerebrovascular history, local anesthetic allergy, opioid allergy, puncture site infection, abnormal clotting.
2. Subjects Patients were allocated randomly to A group (the high fascia iliaca compartment block group) and B group (the femoral nerve block combined with sciatic nerve block group) according to a computer-generated random number table. All patients and an investigator who was responsible for follow-up during 48 postoperative hours were blinded to the randomization groups. In addition, during preoperative visits, the investigators instructed patients on how to use the patient-controlled intravenous analgesia (PCA) device for pain management, as well as how to use the visual analog scale to evaluate pain at rest and while coughing. All the bispectral index (BIS) value in the present study was maintained between 40 and 60 during surgery. All patients voluntarily signed informed consent.
3. General anesthesia Patients were monitored by electrocardiogram, pulse oximetry, and non-invasive blood pressure (one measurement every 3 min) while entering the operation room. A radial artery catheter was also placed for invasive arterial pressure and blood gas monitoring. The induction of general anesthesia was performed intravenously with sufentanil 0.5 µg/kg, propofol 1-2 mg/kg, and rocuronium 0.6 mg/kg. Endotracheal intubation was performed with a double-lumen tube. Sevoflurane was used at a minimal alveolar concentration (MAC) of 0.8-1, remifentanil and propofol were used for the maintenance. Fluid management was at the discretion of the attending anaesthesiologist.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 to 65 years male and female
* Scheduled for elective arthroscopic knee surgery
* The patients volunteered to participate in the study and signed the informed consent

Exclusion Criteria:

* Preexisting neuropathy
* Coagulopathy
* Local skin infection
* Hepatic, renal, or cardiorespiratory failure
* Local anesthetic allergy
* Pregnancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2022-02-05 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-02-05 (Estimated)

PRIMARY OUTCOMES:
The mini-mental State Examination | one day before the operation.
  The mini-mental State Examination is effective as a screening tool for cognitive impairment in older, community-dwelling, hospitalized, and institutionalized adults. Assessment of an older adult's cognitive function is best achieved when it is done routinely, systematically, and thoroughly. The Mini-Mental State Examination (MMSE) or Folstein test is a 30-point questionnaire that is used extensively in clinical and research settings to measure cognitive impairment. Any score of 24 or more (out of 30) indicates normal cognition. Below this, scores can indicate severe (≤9 points), moderate (10-18 points), or mild (19-23 points) cognitive impairment. The raw score may also need to be corrected for educational attainment and age.
Change from Baseline visual analogue scale | 30 minutes after extubation and 6 hours and 12 hours
  Using a ruler, the score is determined by measuring the distance (mm) on the 10-cm line between the "no pain" anchor and the patient's mark, providing a range of scores from 0 to 100. A higher score indicates greater pain intensity. Based on the distribution of pain Visual Analogue Scale scores in post-surgical patients (knee replacement, hysterectomy, or laparoscopic myomectomy) who described their postoperative pain intensity as none, mild, moderate, or severe, the following cut points on the pain Visual Analogue Scale have been recommended: no pain (0-4 mm), mild pain(5-44 mm), moderate pain (45-74 mm), and severe pain (75-100 mm).

SECONDARY OUTCOMES:
The effective times of patient-controlled intravenous analgesia | during 0-6 hours, 6-12 hours, and 12-24 hours
  Change from Baseline patient-controlled intravenous analgesia

CONTACTS AND LOCATIONS:
Overall Officials: Tao Zhang, Principal Investigator — Ethics Committee of Affiliated Hospital of Nantong University
Locations (1):
- Affiliated Hospital of Nantong University, Nantong, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No